CLINICAL TRIAL: NCT04524273
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Phase 3 Study With Open-label Period to Evaluate the Efficacy and Safety of Inebilizumab in Adults With Myasthenia Gravis
Brief Title: Myasthenia Gravis Inebilizumab Trial
Acronym: MINT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIB0551.P3.S1
Expanded Access: NCT06590051 (Available)
Record Dates: First submitted 2020-08-10; First posted 2020-08-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — inebilizumab

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Multicenter, Placebo-controlled Phase 3 Study with Open-label Period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study in which the IV inebilizumab and the IV placebo are matching in appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inebilizumab, (AChR-Ab+) MG (Experimental): Participants will receive inebilizumab administered intravenously (IV) on Days 1, 15, and 183 of the RCP.
  Participants who elect to enter the open label phase (OLP) will receive inebilizumab administered IV on OLP Days 1, IV placebo on OLP Day 15 (to avoid potential unblinding), and inebilizumab IV on OLP Days 183, 365, 547, 729, and 911.
  Interventions: Drug: inebilizumab
- Placebo, (AChR-Ab+) MG (Placebo Comparator): Participants will receive placebo administered IV on Days 1, 15, and 183 of the RCP.
  Participants who elect to enter the OLP will receive inebilizumab administered IV on OLP Days 1,15, 183, 365, 547, 729, and 911.
  Interventions: Drug: IV Placebo
- Inebilizumab, (MuSK-Ab+) MG (Experimental): Participants will receive inebilizumab administered IV on Days 1 and 15 of the RCP.
  Participants who elect to enter the OLP will receive inebilizumab administered IV on OLP Day 1, IV placebo on OLP Day 15 (to avoid potential unblinding), and inebilizumab IV on OLP Days 183, 365, 547, 729, and 911.
  Interventions: Drug: inebilizumab
- Placebo, (MuSK-Ab+) MG (Placebo Comparator): Participants will receive placebo administered IV on Days 1 and 15 of the RCP. Participants who elect to enter the OLP will receive inebilizumab administered IV on OLP Days 1,15, 183, 365, 547, 729, and 911.
  Interventions: Drug: IV Placebo

INTERVENTIONS:
Drug: inebilizumab — Participants will receive IV inebilizumab
  Other Names: MEDI-551; VIB0551
  Arms: Inebilizumab, (AChR-Ab+) MG; Inebilizumab, (MuSK-Ab+) MG
Drug: IV Placebo — Participants will receive IV placebo matched to inebilizumab
  Arms: Placebo, (AChR-Ab+) MG; Placebo, (MuSK-Ab+) MG

SUMMARY:
Randomized, double-blind, placebo-controlled, Phase 3, parallel-group study with optional open-label extension.

DETAILED DESCRIPTION:
This study is a phase 3, randomized, double-blind, placebo-controlled study, to be conducted at approximately 120 study sites. Approximately 230 participants (188 acetylcholine receptor antibody positive [AChR-Ab+] and 42 muscle-specific tyrosine kinase antibody positive [MuSK-Ab+]) will be enrolled. Participants with Myasthenia Gravis (MG) who are positive for anti-AChR or anti-MuSK antibodies will be enrolled and analyzed. Patients who do not have anti-AChR or anti-MuSK antibodies will not be enrolled. Patients with Myasthenia Gravis Foundation of America (MGFA) classification II, III, or IV disease, Myasthenia Gravis Activities of Daily Living (MG-ADL) score at screening and randomization between 6 and 10 with > 50% of this score attributed to non-ocular items, or an MG-ADL score >=11, Quantitative Myasthenia Gravis (QMG) score >= 11 at the time of screening and randomization, and use of a corticosteroid and/or non-steroidal immunosuppressant will be included in the study.

All subjects who complete the randomized controlled period (RCP) will have the option to enroll in a 3-year (156 weeks) open-label period.

Study acquired from Horizon in 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MG with anti-AChR or anti-MuSK antibody.
2. MGFA Clinical Classification Class II, III, or IV.
3. MG-ADL score of 6 or greater at screening and at randomization with > 50% of this score attributed to non-ocular items.
4. QMG score of 11 or greater.
5. Participants must be on:

   1. Corticosteroids only, with no dose increase within 4 weeks prior to randomization, or
   2. One allowed non-steroidal immunosuppressive therapy (IST), with continuous use for at least 6 months prior to randomization and no dose increase within 4 months prior to randomization, or
   3. Combination of (1) corticosteroids with no dose increase within 4 weeks prior to randomization and (2) one allowed non-steroidal IST with continuous use for at least 6 months prior to randomization and no dose increase within 4 months prior to randomization.

Allowed ISTs, alone or in combination with corticosteroids, are azathioprine, mycophenolate mofetil, and mycophenolic acid.

Exclusion Criteria:

1. Receipt of the following medications within the 4 weeks prior to Day 1:

   1. Cyclosporine (except eye drops)
   2. Tacrolimus (except topical)
   3. Methotrexate
2. Current use of:

   1. Corticosteroids (Prednisone > 40 milligram (mg)/day or > 80 mg over a 2-day period (or equivalent dose of other corticosteroids).
   2. Acetylcholinesterase inhibitors (pyridostigmine) > 480 mg/day) or unstable dose in the 2 weeks prior to Day 1.
   3. Azathioprine > 3 mg/kilogram (kg)/day
   4. Mycophenolate mofetil > 3 grams/day or mycophenolic acid > 1440 mg/day
   5. Any IST, alone or in combination with corticosteroids, except for azathioprine, mycophenolate mofetil, and mycophenolic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2027-11-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) Profile score. | Baseline to Week 26

SECONDARY OUTCOMES:
Change from baseline in Quantitative Myasthenia Gravis (QMG) scores. | Baseline to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Proportion of participants with both ≥ 3-point improvement from baseline in MG-ADL and did not initiate rescue therapy. | Baseline to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Change from baseline in MG-ADL | Baseline to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Time to first gMG exacerbation. | Day 1 to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Change from baseline in Myasthenia Gravis Composite (MGC) score. | Baseline to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Change from baseline in Myasthenia Gravis Quality of Life-15, revised (MGQOL-15r) score. | Baseline to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Patient Global Impression of Change (PGIC) score. | Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Number of participants with treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), and treatment-emergent serious adverse events (TESAEs) during the RCP and OLP. | Up to 208 weeks
Proportion of participants with steroid tapered to ≤ 5 mg/day. | Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Proportion of participants with a steroid dose reduction from baseline of ≥ 50%. | Baseline to Week 52 for AChR-Ab+ population and Week 26 for the overall study population
Proportion of participants achieving minimal symptom expression. | Week 26
  Minimal symptom expression was defined as an MG-ADL of 0 or 1.
Proportion of participants with anti-drug antibodies (ADAs) to inebilizumab | Up to 208 weeks
Titers of ADAs | Up to 208 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (104):
- United States (16):
  - Viela Bio Investigative Site - 1015, Orange, California
  - Viela Bio Investigative Site - 1002, New Haven, Connecticut
  - Viela Bio Investigative Center - 1024, Washington D.C., District of Columbia
  - Viela Bio Investigative Site - 1005, Tampa, Florida
  - Viela Bio Investigative Site - 1012, Kansas City, Kansas
  - Viela Bio Investigative Site - 1018, Charlotte, North Carolina
  - Viela Bio Investigative Site - 1025, Canton, Ohio
  - Viela Bio Investigative Site - 1001, Cincinnati, Ohio
  - Viela Bio Investigative Site - 1009, Columbus, Ohio
  - Viela Bio Investigative Site - 1008, Pittsburgh, Pennsylvania
  - Viela Bio Investigative Site - 1019, Austin, Texas
  - Viela Bio Investigative Site - 1003, Houston, Texas
  - Viela Bio Investigative Site - 1014, San Antonio, Texas
  - Viela Bio Investigative Site - 1017, Salt Lake City, Utah
  - Viela Bio Investigative Site - 1004, Burlington, Vermont
  - Viela Bio Investigative Site - 1006, Richmond, Virginia
- Argentina (3):
  - Viela Bio Investigative Site - 2001, Buenos Aires
  - VielaBio Investigative Site - 2002, Buenos Aires
  - Viela Bio Investigative Site - 2003, Buenos Aires
- Belarus (3):
  - Viela Bio Investigative Site - 5203, Grodno
  - Viela Bio Investigative Site - 5204, Minsk
  - Viela Bio Investigative Site - 5201, Vitebsk
- Brazil (5):
  - VielaBio Investigative Site - 2201, Porto Alegre
  - VielaBio Investigative Site - 2203, Porto Alegre
  - VielaBio Investigative Site - 2207, Ribeirão Preto
  - VielaBio Investigative Site - 2206, São Paulo
  - Viela Bio Investigative Site - 2205, São Paulo
- Canada (3):
  - Viela Bio Investigative Site - 1102, Toronto, Ontario
  - Viela Bio Investigative Site - 1101, Montreal, Quebec
  - Viela Bio Investigative Site - 1103, Montreal, Quebec
- China (10):
  - Viela Bio Investigative Site 4009, Beijing
  - Viela Bio Investigative Site - 4007, Beijing
  - Viela Bio Investigative Site 4003, Beijing
  - Viela Bio Investigative Site - 4005, Guiyang
  - Viela Bio Investigative site 4010, Hunan
  - Viela Bio Investigative Site - 4011, Jinan
  - Viela Bio Investigative Site - 4006, Shanghai
  - Viela Bio Investigative Site - 4008, Suzhou
  - Viela Bio Investigative Site - 4004, Tianjin
  - Viela Bio Investigative Site 4012, Xi'an
- Viela Bio Investigative Site - 5601, Copenhagen, Denmark
- France (3):
  - Viela Bio Investigative Site - 3003, Lille
  - Viela Bio Investigative Site - 3001, Nice
  - Viela Bio Investigative Site - 3002, Strasbourg
- VielaBio Investigative Site - 3101, Essen, Germany
- India (9):
  - Viela Bio Investigative Site - 4107, Nagpur, Maharashtra
  - Viela Bio Investigative Site - 4113, Nagpur, Maharashtra
  - Viela Bio Investigative Site - 4112, Hyderabad, Telangana
  - Viela Bio Investigative Site - 4104, Bangalore
  - Viela Bio investigative Site - 4105, Lucknow
  - Viela Bio Investigative Site - 4103, Manipal
  - Viela Bio Investigative Site - 4102, Nashik
  - Viela Bio Investigative Site - 4109, Pune
  - Viela Bio Investigative Site - 4101, Surat
- Italy (4):
  - Viela Bio Investigative Site - 3204, Milan
  - Viela Bio Investigative Site - 3203, Milan
  - Viela Bio Investigative Site - 3201, Pavia
  - Viela Bio Investigative Site - 3202, Rome
- Japan (10):
  - Viela Bio Investigative Site - 4402, Chiba
  - Viela Bio Investigative Site - 4410, Chiba
  - Viela Bio Investigative Site 4409, Fukuoka
  - Viela Bio Investigative Site - 4401, Hanamaki
  - VielaBio Investigative Site - 4408, Hokkaido
  - Viela Bio Investigative Site - 4406, Hyōgo
  - Viela Bio Investigative Site 4405, Miyagi
  - Viela Bio Investigative Site - 4413, Moriguchi
  - VielaBio Investigative Site - 4407, Morioka
  - Viela Bio Investigative Site - 4404, Saitama
- Poland (5):
  - Viela Bio Investigative Site - 3302, Katowice
  - Viela Bio Investigative Site - 3303, Katowice
  - Viela Bio Investigative Site - 3301, Krakow
  - Med Polonia Sp. z o.o - 3311, Poznan
  - Viela Bio Investigative Site - 3310, Warsaw
- Russia (9):
  - Viela Bio Investigative Site - 5313, Barnaul, Altayskiy Kray
  - Viela Bio Investigative Site - 5303, Barnaul
  - Viela Bio Investigative Site - 5302, Nizhny Novgorod
  - Viela Bio Investigative Site - 5304, Novosibirsk
  - Viela Bio Investigative Site - 5311, Rostov-on-Don
  - Viela Bio Investigative Site - 5309, Rostov-on-Don
  - Viela Bio Investigative Site - 5308, Saint Petersburg
  - Viela Bio Investigative Site - 5305, Samara
  - Viela Bio Investigative Site - 5312, Ufa
- South Korea (3):
  - Viela Bio Investigative Site - 4202, Seoul
  - Viela Bio Investigative Site - 4203, Seoul
  - Viela Bio Investigative Site - 4201, Seoul
- Spain (3):
  - Viela Bio Investigative Site - 3403, Badalona
  - Viela Bio Investigative Site - 3402, Barcelona
  - Viela Bio Investigative Site - 3404, Córdoba
- Taiwan (7):
  - Viela Bio investigative Site - 4605, Kaohsiung City
  - Viela Bio Investigative Site 4608, New Taipei City
  - Viela Bio Investigative Site - 4606, Tainan
  - Viela Bio Investigative Site - 4604, Taipei
  - Viela Bio Investigative Site - 4603, Taipei
  - Viela Bio Investigative Site -4607, Taipei
  - Viela Bio Investigative Site - 4602, Taoyuan
- Turkey (Türkiye) (4):
  - Viela Bio Investigative Site - 3903, Ankara
  - Viela Bio Investigative Site - 3901, Izmir
  - Viela Bio Investigative Site - 3902, Izmir
  - Viela Bio Investigative Site - 3905, Kocaeli
- Ukraine (5):
  - Viela Bio Investigative Site - 5103, Dnipro
  - Viela Bio Investigative Site - 5108, Dnipro
  - Viela Bio Investigative Site - 5105, Ivano-Frankivsk
  - Viela Bio Investigative Site - 5104, Lutsk
  - Viela Bio Investigative Site - 5106, Vinnytsia

REFERENCES:
- [Derived] Nowak RJ, Benatar M, Ciafaloni E, Howard JF Jr, Leite MI, Utsugisawa K, Vissing J, Rojavin M, Li Q, Tang F, Wu Y, Rampal N, Cheng S; MINT Investigators. A Phase 3 Trial of Inebilizumab in Generalized Myasthenia Gravis. N Engl J Med. 2025 Jun 19;392(23):2309-2320. doi: 10.1056/NEJMoa2501561. Epub 2025 Apr 8. PMID 40202593
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com